CLINICAL TRIAL: NCT05063942
Title: Does Covid-19 Vaccination in Patients Undergoing in Vitro Fertilization Affect the Live Birth Rate of Their First Embryo Transfer Cycle: A Prospective Cohort Study
Brief Title: The Effect of Covid-19 Vaccination in Patients Undergoing IVF
Acronym: Covid-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, chen zhi qin, Professor, Shanghai First Maternity and Infant Hospital
Other Study IDs: 001
Record Dates: First submitted 2021-09-30; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Covid-19 Vaccination
Keywords: IVF Covid-19 Vaccination live birth rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since emerging in the last months of 2019, over 127 000 000 individuals have suffered severe acute respiratory syndrome Coronavirus 2 (SARS-CoV-2) infection, and the documented death toll from coronavirus disease 2019 (COVID-19) had reached 2788639 individuals globally by the end of March 2021 (CDC, 2021).It is hoped that widespread vaccination will further limit viral spread and shorten the length of the pandemic and its impact on morbidity and mortality. There are currently two vaccines against the new coronavirus: inactivated vaccines and mRNA vaccines.Nationwide anti-COVID-19 vaccination began in China in March 2020, using the inactivated vaccine. By the end of September 2021, 2206.054 million doses (including the first and second doses of the vaccine) of the vaccines have been fulfilled.There is still a lack of real-world data to assist clinicians in counseling their IVF patients regarding the possible impact of recent recovery from COVID infection, or vaccination against it, on the potential for success of ART. We aimed to determine the impact of confirmed COVID-19 immunization on IVF outcomes, by comparing live birth rate of the first transfer cycle in patients undergoing IVF with and without COVID- 19 vaccination.

DETAILED DESCRIPTION:
Since emerging in the last months of 2019, over 127 000 000 individuals have suffered severe acute respiratory syndrome Coronavirus 2 (SARS-CoV-2) infection, and the documented death toll from coronavirus disease 2019 (COVID-19) had reached 2788639 individuals globally by the end of March 2021 (CDC, 2021).Although a major victory has been achieved in the fight against the epidemic since first case was reported in Wuhan City,, the cumulative death toll is 5,691 by the end of September in China . At the present time, mitigation strategies for controlling the pandemic continue to rely heavily on universal masking, physical distancing, limiting social interactions, and frequent sanitizing measures. It is hoped that widespread vaccination will further limit viral spread and shorten the length of the pandemic and its impact on morbidity and mortality.

There are currently two vaccines against the new coronavirus: inactivated vaccines and mRNA vaccines. Unlike inactivated vaccines, the mRNA vaccine does not use natural pathogens, but artificially synthesizes the gene sequence encoding a specific antigen protein, and then directly injects the mRNA encoding the antigen protein into the human body to induce the immune system to produce antibodies against the new coronavirus. Although some studies have shown that mRNA vaccines do not increase the risk of miscarriage in women, the conclusion is limited due to the lack of non-pregnant women as a control group. At the same time, the impact of inactivated vaccines on female pregnancy is still in a blank state. Nationwide anti-COVID-19 vaccination began in China in March 2020, using the inactivated vaccine vaccine. By the end of September 2021, 2206.054 million doses (including the first and second doses of the vaccine) of the vaccines have been fulfilled. We aimed to determine the impact of confirmed COVID-19 immunization on IVF outcomes, by comparing live birth rate of the first transfer cycle in patients undergoing IVF with and without COVID- 19 vaccination.

ELIGIBILITY:
Inclusion Criteria:

Age of women <43 years at the time of ovarian stimulation for IVF

Exclusion Criteria:

1. an abnormal uterine cavity shown on hysterosalpingogram or hysteroscopy,
2. moderate or severe endometriosis,
3. Recipient of oocyte donation and
4. Undergoing preimplantation genetic testing
5. Presence of hydrosalpinx or endometrial polyp which is not surgically treated
6. patients with poor ovarian response (less than 3 mature follicles)

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing IVF with and without COVID- 19 vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 712 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
live birth rate per transfer | 10 month
  A baby born alive after 22 weeks gestation was classified as a live birth

SECONDARY OUTCOMES:
biochemical pregnancy rate | 2 weeks
  positive urine pregnancy test
clinical pregnancy rate | 4 weeks
  presence of intrauterine gestational sac on ultrasound
embryo implantation rate | 2month
  number of gestational sacs per embryo transferred
number of transferable embryos | 2weeks
  Number of oocytes retrieved and embryos/blastocysts suitable for freezing and transfer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Esposito V, Rania E, Lico D, Pedri S, Fiorenza A, Strati MF, Conforti A, Marrone V, Carosso A, Revelli A, Zullo F, Di Carlo C, Venturella R. Influence of COVID-19 pandemic on the psychological status of infertile couples. Eur J Obstet Gynecol Reprod Biol. 2020 Oct;253:148-153. doi: 10.1016/j.ejogrb.2020.08.025. Epub 2020 Aug 23. PMID 32866858
- [Result] Abu Jabal K, Ben-Amram H, Beiruti K, Batheesh Y, Sussan C, Zarka S, Edelstein M. Impact of age, ethnicity, sex and prior infection status on immunogenicity following a single dose of the BNT162b2 mRNA COVID-19 vaccine: real-world evidence from healthcare workers, Israel, December 2020 to January 2021. Euro Surveill. 2021 Feb;26(6):2100096. doi: 10.2807/1560-7917.ES.2021.26.6.2100096. PMID 33573712
- [Result] Jing Y, Run-Qian L, Hao-Ran W, Hao-Ran C, Ya-Bin L, Yang G, Fei C. Potential influence of COVID-19/ACE2 on the female reproductive system. Mol Hum Reprod. 2020 Jun 1;26(6):367-373. doi: 10.1093/molehr/gaaa030. PMID 32365180
- [Result] Zambrano LD, Ellington S, Strid P, Galang RR, Oduyebo T, Tong VT, Woodworth KR, Nahabedian JF 3rd, Azziz-Baumgartner E, Gilboa SM, Meaney-Delman D; CDC COVID-19 Response Pregnancy and Infant Linked Outcomes Team. Update: Characteristics of Symptomatic Women of Reproductive Age with Laboratory-Confirmed SARS-CoV-2 Infection by Pregnancy Status - United States, January 22-October 3, 2020. MMWR Morb Mortal Wkly Rep. 2020 Nov 6;69(44):1641-1647. doi: 10.15585/mmwr.mm6944e3. PMID 33151921
- See also: Vaccinating pregnant and lactating patients against COVID-19 — http://www.acog.org/clinical/clinical-guidance/practice-advisory/articles/2020/12/covid-19-vaccination-considerations-for-obstetric-gynecologic-care?utm_source=redirect&utm_medium=web&utm_campaign=int